CLINICAL TRIAL: NCT02059590
Title: A Phase 1 Open-Label Mass Balance Study to Evaluate the Pharmacokinetics of BAL8728 After A Single Intravenous Dose of 14C-Labeled Isavuconazonium Sulfate in Healthy Male Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics of BAL8728 After a Single Dose of Pyridinylmethyl-14C-Labeled Isavuconazonium Sulfate in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0050
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Pharmacokinetics of 14C-labeled Isavuconazonium Sulfate; Healthy Subjects
Keywords: 14C-labeled isavuconazonium sulfate; Pyridinylmethyl-14C-labeled isavuconazonium sulfate; Healthy Subjects; BAL8728; BAL4815
MeSH Terms: interventions — isavuconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pyridinylmethyl-14C-labeled isavuconazonium sulfate (Experimental): single dose
  Interventions: Drug: Pyridinylmethyl-14C-labeled isavuconazonium sulfate

INTERVENTIONS:
Drug: Pyridinylmethyl-14C-labeled isavuconazonium sulfate — Intravenous
  Other Names: BAL8557

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of 14C-labeled cleavage product (BAL8728), in particular the routes of excretion and extent ot metabolism of the cleavage product following administration of a single intravenous dose of pyridinylmethyl-14C-labeled prodrug isavuconazonium sulfate (BAL8557). In addition, identify the metabolic profile of BAL8728 in human plasma, urine and/or feces after a single intravenous dose of pyridinylmethyl-14C-labeled BAL8557 and evaluate the pharmacokinetics of BAL8728 and BAL4815. Safety and tolerability after a single intravenous dose of pyridinylmethyl-14C-labeled isavuconazonium sulfate will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45 kg and a body mass index of 18 to 32 kg/m2, inclusive.
* The subject's 12-lead electrocardiogram (ECG) is normal at Screening and Day -1; or, if abnormal, the abnormality is not clinically significant. The ECG for the subject has a QTcF of at least 360 but not more than 430 msec.

Exclusion Criteria:

* The subject has any clinically significant disease history of the following systems: pulmonary, gastrointestinal, cardiovascular (including a history of clinically significant arrhythmia), hepatic, neurological, psychiatric, renal, genitourinary, endocrine, metabolic, dermatologic, immunologic, hematologic, or malignancy excluding non melanoma skin cancer.
* The subject has a positive test for hepatitis B surface antigen or hepatitis C antibodies at Screening or is known to be positive for human immunodeficiency virus.
* The subject has a known or suspected allergy to any of the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reactions.
* The subject has used tobacco or nicotine containing products in the last 6 months prior to Day -1.
* The subject has had treatment with prescription drugs, over-the-counter medication, or complementary and alternative medicines within 14 days prior to Day -1, with the exception of occasional use of acetaminophen up to 2 g/day.
* The subject has participated in any interventional clinical study or has received any investigational agent within 28 days or 5 half-lives, whichever is longer, prior to Screening.
* The subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission on Day -1.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Radioactivity in whole blood and in plasma: Area under the concentration-time curve (AUC) from time of dosing to infinity (AUCinf) | 20 time points up to Day 4. If Day 4 is not the end of the study, samples will be drawn once a day up to Day 9
Radioactivity in whole blood and in plasma: AUC from time of dosing to the last quantifiable concentration (AUClast) | 20 time points up to Day 4. If Day 4 is not the end of the study, samples will be drawn once a day up to Day 9
Radioactivity in whole blood and in plasma: Maximum concentration (Cmax) | 20 time points up to Day 4. If Day 4 is not the end of the study, samples will be drawn once a day up to Day 9
Radioactivity in whole blood and in plasma: Time to Attain Cmax (tmax) | 20 time points up to Day 4. If Day 4 is not the end of the study, samples will be drawn once a day up to Day 9
Radioactivity in whole blood and in plasma: Apparent terminal elimination half-life (t1/2) | 20 time points up to Day 4. If Day 4 is not the end of the study, samples will be drawn once a day up to Day 9
Radioactivity in emesis (if applicable) | After study drug administration up to Day 9
Radioactivity ratio blood/plasma | Day 1
Percent of dose and cumulative percent of dose of radioactivity recovered in urine | 7 time intervals up to Day 4. If Day 4 is not the end of the study, sample collection will continue in 24 hour intervals until discharge up to Day 9
Percent of dose and cumulative percent dose of radioactivity recovered in feces | 4 time intervals up to Day 4. If Day 4 is not the end of the study, sample collection will continue in 24 hour intervals until discharge up to Day 9
Pharmacokinetics of BAL8728 (cleavage product) in plasma: AUCinf | 20 time points up to Day 4. If Day 4 is not the end of the study, samples will be drawn once a day up to Day 9
Pharmacokinetics of BAL8728 (cleavage product) in plasma: AUClast | 20 time points up to Day 4. If Day 4 is not the end of the study, samples will be drawn once a day up to Day 9
Pharmacokinetics of BAL8728 (cleavage product) in plasma: Cmax | 20 time points up to Day 4. If Day 4 is not the end of the study, samples will be drawn once a day up to Day 9
Pharmacokinetics of BAL8728 (cleavage product) in plasma: tmax | 20 time points up to Day 4. If Day 4 is not the end of the study, samples will be drawn once a day up to Day 9
Pharmacokinetics of BAL8728 (cleavage product) in plasma: total body clearance after intravenous dosing (CLtot) | 20 time points up to Day 4. If Day 4 is not the end of the study, samples will be drawn once a day up to Day 9
Pharmacokinetics of BAL8728 (cleavage product) in plasma: volume of distribution during terminal phase after intravenous dosing (Vz) | 20 time points up to Day 4. If Day 4 is not the end of the study, samples will be drawn once a day up to Day 9
Pharmacokinetics of BAL8728 (cleavage product) in plasma: t 1/2 | 20 time points up to Day 4. If Day 4 is not the end of the study, samples will be drawn once a day up to Day 9
Pharmacokinetics of BAL8728 (cleavage product) in urine: amount excreted (Ae) | 7 time intervals up to Day 4. If Day 4 is not the end of the study, sample collection will continue in 24 hour intervals until discharge up to Day 9
Pharmacokinetics of BAL8728 (cleavage product) in urine: percent of unchanged drug excreted into the urine (Ae%) | 7 time intervals up to Day 4. If Day 4 is not the end of the study, sample collection will continue in 24 hour intervals until discharge up to Day 9
Pharmacokinetics of BAL8728 (cleavage product) in urine: renal clearance (CLr) | 7 time intervals up to Day 4. If Day 4 is not the end of the study, sample collection will continue in 24 hour intervals until discharge up to Day 9
Pharmacokinetics of BAL4815 (isavuconazole) in plasma: AUClast | 20 time points up to Day 4. If Day 4 is not the end of the study, samples will be drawn once a day up to Day 9
Pharmacokinetics of BAL4815 (isavuconazole) in plasma: Cmax | 20 time points up to Day 4. If Day 4 is not the end of the study, samples will be drawn once a day up to Day 9
Pharmacokinetics of BAL4815 (isavuconazole) in plasma: tmax | 20 time points up to Day 4. If Day 4 is not the end of the study, samples will be drawn once a day up to Day 9

SECONDARY OUTCOMES:
Metabolic profile of BAL8728 and possible metabolites in plasma, urine, and feces | Up to 3 days (72 hours) after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Covance, Madison, Wisconsin, United States